CLINICAL TRIAL: NCT05066893
Title: Type 1 Diabetes Boot Camp Program: An Intensive Program to Improve Glycemic Control in Adolescents With Type 1 Diabetes
Brief Title: Pediatric Boot Camp Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2604
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Type 1 Diabetes; Children, Only
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (Active Comparator): standard of care will be given as per usual care
  Interventions: Other: telehealth visits
- intensive monitoring (Experimental): intensive monitoring every week will be given to participants
  Interventions: Other: telehealth visits

INTERVENTIONS:
Other: telehealth visits — intensive visits with doctor

SUMMARY:
An intensive 13 weeks program that aims to improve glucose control in children with type 1 diabetes.

DETAILED DESCRIPTION:
Our new PeDi-BoCa Program aims to help children with type 1 diabetes achieve better diabetes control by interacting weekly with their doctor/nurse practitioner (NP) and also by using a "smart pen" that can facilitate the burden of daily calculations with the use of an app on the phone.

Your child's doctor/NP will be able to remotely monitor your child's glucose every week (Dexcom) and make recommendations for changes, discuss solutions to possible obstacles and offer intensive diabetes education.

ELIGIBILITY:
Inclusion Criteria:

1. Age 11-18 years old
2. HbA1c > 8.5%
3. Duration of type 1 diabetes >1 year
4. Child uses Dexcom and has a phone that is compatible with the InPen app and Dexcom Clarity app.

Exclusion Criteria:

Not able to attend telehealth visits

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-11-05 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medstar Pediatrics, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No